CLINICAL TRIAL: NCT04403113
Title: The Effects of Neurodevelopmental Therapy on Feeding and Swallowing Activities in Children With Cerebral Palsy.
Brief Title: The Effects of Neurodevelopmental Therapy on Feeding and Swallowing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09.2018.278
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Cerebral Palsy
Keywords: Neck-trunk stabilization exercise. Feeding. Swallowing
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (SG) (Experimental): feeding and oral motor intervention strategies+structured neck and trunk stabilization exercises+caregiver training related to feeding (Study Group)
  Interventions: Other: Structured neck and trunk stabilization exercises; Other: Feeding and oral motor intervention strategies; Other: Caregiver training related to feeding
- Control Group (CG). (Placebo Comparator): feeding and oral motor intervention strategies+caregiver training related to feeding (Control Group)
  Interventions: Other: Feeding and oral motor intervention strategies; Other: Caregiver training related to feeding

INTERVENTIONS:
Other: Structured neck and trunk stabilization exercises — Intensive structured neck and trunk stabilization exercises based on Neurodevelopmental therapy method-Bobath concept principles. These exercises were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
  Arms: Study Group (SG)
Other: Feeding and oral motor intervention strategies — Feeding and oral motor intervention strategies program were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
Other: Caregiver training related to feeding — In caregiver training related to feeding; a) positioning and feeding technique during feeding, b) ensuring safety for aspiration, c) using suitable containers and ingredients, d) adjusting (adapting) food consistency properly, e) preparing small amounts of high-calorie, balanced diet and f) reducing food spillage while feeding and how to ensure efficacy for shortening the feeding time, g) providing appropriate postural and physical support for self-feeding. All of these activities were continued for 6 weeks with a home program.

SUMMARY:
Our study is planned to investigate the effects of neck and trunk stabilization exercises, which are structured from Neurodevelopmental therapy method-Bobath concept (NDT-B) principles, on feeding and swallowing activity in children with Cerebral Palsy (CP) who take feeding and oral motor intervention strategies. The cases were divided into two groups, which is the group receiving feeding and oral motor intervention strategies+structured neck and trunk stabilization exercises (n=20) (Study Group) and those receiving feeding and oral motor intervention strategies (n=20) (Control Group).

DETAILED DESCRIPTION:
Feeding and oral motor interventions address different aspects of feeding difficulties, reflecting the range in specific problems associated with feeding and nutrition in CP.

The trunk plays an important role in the organization of postural control and balance reactions because it holds the centre of all body mass and holds therefore, the centre of gravity. The trunk also provides stable attachment points to those muscles that control the head and neck regions. "Neck and trunk stabilization exercises" were the basis of static and dynamic balance abilities, and that increased neck and trunk stability might have had a positive effect thereon.

To achieve the alignment of the head with the trunk, the pelvis must be stabilized. This has important consequences for the entire process of swallowing. If the head is not stable, then the fine movements of the jaw and tongue needed for feeding will be impaired. With feeding and oral motor interventions and structured neck and trunk stabilization exercises, these parameters are positively affected.

ELIGIBILITY:
Inclusion Criteria:

* Cases with Cerebral Palsy who had difficulties in feeding/swallowing skills.
* Cases who were cooperative without communication barriers and volunteering to participate in the study were included.

Exclusion Criteria:

* In the Videoendoscopic Swallowing Study, he/she was not included in the study if he/she had an aspiration or aspiration risk, had advanced vision and hearing loss, used any pharmacological agent to inhibit spasticity, or had undergone orthopaedic surgery or Botulinum Toxin-A injection in the past six months.

Ages: 18 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasim EJRAEI, Master D, Principal Investigator — Marmara University; Gonul Acar, Assoc. Prof, Study Director — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acar G, Ejraei N, Turkdogan D, Enver N, Ozturk G, Aktas G. The Effects of Neurodevelopmental Therapy on Feeding and Swallowing Activities in Children with Cerebral Palsy. Dysphagia. 2022 Aug;37(4):800-811. doi: 10.1007/s00455-021-10329-w. Epub 2021 Jun 25. PMID 34173063
- See also: Feeding children with cerebral palsy and swallowing difficulties — https://www.nature.com/articles/ejcn2013224#citeas
- See also: The importance of postural control for feeding. — https://www.ncbi.nlm.nih.gov/pubmed/15185730
- See also: The effects of neck and trunk stabilization exercises on cerebral palsy children's static and dynamic trunk balance: case series — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5430291/
- See also: The objective rating of oral-motor functions during feeding — https://link.springer.com/article/10.1007/BF00260975

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group (SG): feeding and oral motor intervention strategies+structured neck and trunk stabilization exercises+caregiver training related to feeding.
  Structured neck and trunk stabilization exercises: Intensive structured neck and trunk stabilization exercises based on Neurodevelopmental therapy method-Bobath concept principles. These exercises were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
  Feeding and oral motor intervention strategies: Feeding and oral motor intervention strategies program were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
  Caregiver training related to feeding: In caregiver training related to feeding; a) positioning and feeding technique during feeding, b) ensuring safety for aspiration, c) using suitable containers and ingredients, d) adjusting (adapting) food consistency properly, e) preparing small amounts of high-calorie, balanced diet and f) reducing food spillage while feeding and how to
Period: Overall Study
Arm/Group | Study Group (SG) | Control Group (CG).
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group (SG) | Control Group (CG). | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Count of Participants; unit: Participants]
  Age range: (18-48 months) < | 13 | 14 | 27
  Age range: ≥ (48 months) | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 8 | 11 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 20 | 19 | 39
  Syria | 0 | 1 | 1
Cerebral Palsy type [Count of Participants; unit: Participants]
  diplegic | 3 | 1 | 4
  hemiplegic | 2 | 2 | 4
  quadriplegic | 8 | 10 | 18
  hypotonic | 6 | 5 | 11
  dyskinetic | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Gross Motor Function Classification System (GMFCS)
Description: The gross motor functions of children with cerebral palsy were classified with GMFCS. GMFCS is a 5-level classification system. It uses gross motor skills. The aim is to present an idea of how self-sufficient a child can be at home, at school, and outdoor and indoor venues. GMFCS includes levels that reflect abilities ranging from unlimited walking (level I) to severe head and trunk control limitations. Requires extensive use of assisted technology and physical assistance, and wheelchair (level V). The higher level in GMFCS means a worse and severe outcome. The low levels mean good motor function.
Time Frame: Immediately before the intervention, the evaluation was performed in the first session (only one time).
Measure: Count of Participants; unit: Participants
Groups:
- Study Group (SG): feeding and oral motor intervention strategies+structured neck and trunk stabilization exercises+caregiver training related to feeding.
  Structured neck and trunk stabilization exercises: Intensive structured neck and trunk stabilization exercises based on Neurodevelopmental therapy method-Bobath concept principles. These exercises were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
  Feeding and oral motor intervention strategies: Feeding and oral motor intervention strategies program were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
  Caregiver training related to feeding.
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
Participants
  level 1 | 4 | 2
  level 2 | 0 | 0
  level 3 | 2 | 0
  level 4 | 4 | 4
  level 5 | 10 | 14

2. Primary Outcome: the Eating and Drinking Ability Classification System (EDACS)
Description: EDACS describes the eating and drinking skills of children with cerebral palsy from the age of 3. It is an ordered scale that defines the degree of assistance required during the meal and the individual's ability to eat and drink between five levels. Level I, safely and efficiently eating and drinking; at level V, it indicates unable to eat or drink safely, relies on tube feeding and is at high risk for aspiration.
Time Frame: Immediately before the intervention, the evaluation was performed in the first session (only one time).
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 16 | 11
Participants
  level 1 | 1 | 0
  level 2 | 3 | 1
  level 3 | 5 | 7
  level 4 | 5 | 2
  level 5 | 2 | 1

3. Primary Outcome: the Mini-Manual Ability Classification System (Mini-MACS)
Description: Mini-MACS is a functional classification that defines how children with cerebral palsy between the ages of 1 and 4 use their hands while holding objects in daily activities. Skill classes at five levels, based on the need for self-help and adaptation when children hold objects. Level I. Handles objects easily and successfully. Level V. Does not handle objects and has severely limited ability to perform even simple actions.
Time Frame: Immediately before the intervention, the evaluation was performed in the first session (only one time).
Measure: Count of Participants; unit: Participants
Groups:
- Study Group (SG): feeding and oral motor intervention strategies+structured neck and trunk stabilization exercises+caregiver training related to feeding
  Structured neck and trunk stabilization exercises: Intensive structured neck and trunk stabilization exercises based on Neurodevelopmental therapy method-Bobath concept principles. These exercises were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
  Feeding and oral motor intervention strategies: Feeding and oral motor intervention strategies program were performed for 6 weeks, 2 days a week, 45 minutes for a total of 12 sessions.
  Caregiver training related to feeding.
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
Participants
  level 1 | 1 | 1
  level 2 | 4 | 3
  level 3 | 5 | 5
  level 4 | 3 | 2
  level 5 | 7 | 9

4. Primary Outcome: Trunk Impairment Scale (TIS)
Description: TIS is a validated scale for cerebral palsy that evaluates the trunk functionally in terms of strength in a sitting position. It also complies with the International Classification of Functionality, Disability and Health in terms of evaluating the static and dynamic balance and trunk coordination of the trunk and the relationship between body function and structures. TIS consists of three subscales: static, dynamic and coordination. For each item; sequential scales with 2, 3 or 4 values are used. The highest scores that can be obtained from the static, dynamic and coordination subscales are; it is 7, 10 and 6 points. Total points are obtained by adding all subscales. The total TIS score ranges from 0 to 23. A high score indicates good trunk control.
Time Frame: Change from TIS was assessed in 0 week (Baseline, in the first session), 6. week (6 weeks after treatment, in the 12th session).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
score on a scale | 5.65 (6.11) | 2.90 (5.28)

5. Primary Outcome: Schedule for Oral Motor Assessment (SOMA)
Description: SOMA is a measure which identifies "oral-motor dysfunction" (OMD). SOMA involves videotaping children and later assessing their feeding skills. Test was implemented in the presence of the child's main caregiver. The entire assessment lasted 20-30 minutes. SOMA has 7 subcategories. Each subcategory has its own cut-off point. Among the "yes" or "no" options opposite the observed parameters, the appropriate one is marked. In some options, the "yes" option indicates an abnormal function, while in some options the "no" option indicates the presence of an abnormal function. BOTTLE, TRAINER CUP, CUP(Cutting Score): ≥ 5 indicates OMD. < 5 indicates normal oral-motor function(OMF). PUREE: ≥ 3 indicates OMD. < 3 indicates normal OMF. SEMI-SOLIDS, SOLIDS: ≥ 4 indicates OMD. < 4 indicates normal OMF. CRACKER: ≥ 9 indicates OMD. < 9 indicates normal OMF. BOTTLE, CUP, PUREE, SOLIDS; minimum(mi) score: 0, maximum(ma): 9. TRAINER CUP; mi: 0, ma: 14. SEMI-SOLIDS; mi: 0, ma: 8. CRACKER; mi: 0, ma: 22.
Time Frame: Change from SOMA was assessed in 0 week (Baseline, in the first session, Before treatment), 6. week (6 weeks after treatment, in the 12th session, After treatment).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (CG). | Study Group (SG)
Number analyzed (Participants) | 20 | 20
score on a scale
  Trainer cup (Before treatment) | 2.10 (1.44) | 3.70 (0.92)
  Trainer cup (After treatment) | 3.75 (1.01) | 3.10 (1.51)
  Puree (Before treatment) | 2.05 (0.99) | 2.10 (1.16)
  Puree (After treatment) | 1.75 (1.20) | 1.55 (1.23)
  Bottle (Before treatment) | 3.55 (1.14) | 2.75 (1.58)
  Bottle (After treatment) | 2.35 (1.63) | 2.70 (1.62)
  Cup (Before treatment) | 2.60 (1.53) | 2.50 (1.57)
  Cup (After treatment) | 2.10 (1.41) | 1.95 (1.53)
  Semi solids (Before treatment) | 2.15 (1.30) | 2.05 (1.39)
  Semi solids (After treatment) | 1.95 (1.39) | 1.90 (1.37)
  Solids (Before treatment) | 2.70 (1.12) | 2.35 (1.42)
  Solids (After treatment) | 2.35 (1.38) | 2.35 (1.38)
  Cracker (Before treatment) | 2.45 (1.31) | 2.25 (1.51)
  Cracker (After treatment) | 2.30 (1.38) | 2.10 (1.37)

6. Primary Outcome: Pediatric Quality of Life Inventory (PedsQL)
Description: The Quality of Life Scale for Children is a general quality of life scale which assesses the physical and psychosocial experiences independent of disease in children between the ages of 2 and 18 years. The scale is composed of 23 items. The items are scored between 0 and 100. The higher the score for the Quality of Life Scale for children, the better is the perception of health-related quality of life. In our study, the total score of the scale was used.
Time Frame: Change from PedsQL was assessed in 0 week (Baseline, in the first session), 6. week (6 weeks after treatment, in the 12th session).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 20 | 20
score on a scale | 48.42 (18.33) | 53.48 (20.28)

7. Other Pre Specified Outcome: Fiberoptic Endoscopic Evaluation of Swallowing (FEES)
Description: Instrumental evaluation of swallowing is a technique that allows the evaluation of swallowing physiology and anatomy in patients. The most commonly used form in the clinic is Flexible Fiberoptic Endoscopic Methods. The structures and functions related to swallowing are evaluated using through a fiberoptic tube extending from the nose to the pharynx. FEES allows direct visualization of some aspects of the pharyngeal phase. It gives information about the physiological changes that occur before and after swallowing. Since velopharyngeal closure occurs during swallowing, observation cannot be made. The pharynx, tongue root vallecula, pyriform sinuses, and residues formed after swallowing in the airway can be traced. There is no uniform decision to decide if a child should switch from oral feeding to enteral tube feeding, but there is a general consensus.
Time Frame: It was applied after the evaluation in the first session.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group (SG) | Control Group (CG).
Number analyzed (Participants) | 4 | 4
Participants
  Normal swallowing and oral diet | 4 | 3
  Dysphagia and non-oral diet | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 weeks for each participant.
Arm/Group | Study Group (SG) | Control Group (CG).
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
In the study, it can be stated as the limitation of the study that all children with feeing problems are screened for only 40 cases and heterogeneous types are included in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT04403113/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT04403113/SAP_001.pdf
  • Informed Consent Form (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT04403113/ICF_002.pdf